CLINICAL TRIAL: NCT02036528
Title: A Phase I/II, Open Label, Controlled Study to Evaluate the Safety and Efficacy of AppliGel-G [Gentamicin Sulfate Topical Gel] for Treatment of Mild to Moderately Infected Diabetic Foot Ulcers in Patients With Type 1 and Type 2 Diabetes
Brief Title: Safety and Efficacy of Gentamicin Topical Gel (AppliGel-G) for Treatment of Mild to Moderately Infected Diabetic Foot Ulcers
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Royer Biomedical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP-RBM-2011-001 DFU
Record Dates: First submitted 2014-01-10; First posted 2014-01-15 (Estimated); Last update posted 2015-05-14 (Estimated); Status verified 2015-05

CONDITIONS: Diabetic Foot Ulcers
Keywords: Foot Ulcer; Diabetic Foot; Gentamicins; infection
MeSH Terms: conditions — Diabetic Foot; Foot Ulcer; Infections | interventions — Ciprofloxacin; Doxycycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AppliGel-G with oral Ciprofloxacin and Doxycycline (Experimental): AppliGel-G (Gentamicin Topical Gel) in conjunction with oral Ciprofloxacin and Doxycycline
  Interventions: Drug: Gentamicin Topical Gel; Drug: Ciprofloxacin; Drug: Doxycycline
- Oral Ciprofloxacin and Doxycycline only (Active Comparator): Ciprofloxacin and Doxycycline
  Interventions: Drug: Ciprofloxacin; Drug: Doxycycline

INTERVENTIONS:
Drug: Gentamicin Topical Gel
  Arms: AppliGel-G with oral Ciprofloxacin and Doxycycline
Drug: Ciprofloxacin
Drug: Doxycycline

SUMMARY:
The purpose of this study is to determine whether AppliGel-G (Gentamicin topical gel) plus oral Ciprofloxacin / Doxycycline are safe and effective in the treatment of mild to moderately infected foot ulcers in diabetic patients.

DETAILED DESCRIPTION:
Infection of a diabetic foot ulcer (DFU) is a serious and common complication of diabetes and is among the most common diabetes-related cause of hospitalization and the leading cause of diabetes-associated lower limb amputation. The effectiveness of various systemic antibiotics, particularly the fluoroquinolones, in treating infected DFUs has been demonstrated.

An alternative or adjunct to systemic antibiotic treatment of infected DFU's is topical antibiotic treatment. Topical treatment would have the advantages of avoiding systemic adverse effects, providing increased target site concentration, and allowing the use of antibiotics not approved for systemic treatment.

AppliGel-G is a topically applied hydrogel formulation of gentamicin sulfate (GMS). Once in place the product remains in contact with the wound bed and releases Gentamicin to the wound bed.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 18 years of age or older
2. Subject has a mild to moderately infected (IDSA Mild or Moderate/ PEDIS Grade 2 or 3) diabetic foot ulcer and without a previous history of partial foot amputation.
3. Subject has Diabetes Mellitus (type 1 or type 2).
4. Wound area measurement between 1-25 cm2 and does not exceed 25 cm2.
5. Subject is in general good health in the opinion of the investigator as determined by medical history, vital signs and a physical examination.
6. Female subjects must have a negative urine pregnancy test at screening and be willing and able to use a medically acceptable method of birth control or declare that they are abstaining from sexual intercourse, from the screening visit through the study termination visit or be surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy) or post-menopausal. Postmenopausal women are defined as women with menstruation cessation for 12 consecutive months prior to signing of the informed consent form.
7. Subject has either no renal failure or only mild renal failure (i.e.: glomerular filtration rate (GFR) must be above 60 mL/min/1.73m2)
8. Subject is willing and committed to comply with the research protocol and complete all outcome measures.
9. Subject is able to self-consent.
10. Subject is able to speak and read English..

Exclusion Criteria:

1. Subject is non-diabetic
2. Subject's foot lesion(s) are of etiology other than diabetic neuropathy
3. DFU is PEDIS Infection Grade 1 or 4
4. Infected DFU measures >25 cm2
5. The wound involves bone, tendon or joint damage not due to infection
6. Wound with sinus tracts
7. HbA1c>11%
8. Subject with skin disorders unrelated to the ulcer that are presented adjacent to the wound
9. Clinically significant arterial vascular disease based on Skin Perfusion Pressure System (SensiLase) measurement of skin perfusion pressure (SPP) of <30 mm Hg.
10. Subject is receiving, or has received within one month prior to enrollment any treatment known to impair wound healing, including but not limited to: corticosteroids, immuno-suppressive drugs, cytotoxic agents, radiation therapy and chemotherapy.
11. Known history of a significant medical disorder, which in the investigator's judgment contraindicates the subject's participation.
12. Has active malignant disease of any kind. A subject, who has had a malignant disease in the past, was treated and is currently disease-free, may be considered for study entry.
13. Subjects who present with significant metabolic co morbidity that would preclude wound healing such as end stage renal failure, dialysis or severe liver dysfunction.
14. Known hypersensitivity and/or allergy to gentamicin or the study oral antibiotics or related drugs.
15. Drug or alcohol abuse (by history). 16 Subjects participating in any other trials in regards to the diabetic foot ulcer or antibiotic therapy.

17 History of myasthenia gravis 18 Any condition or use of prescribed medication in which participation in this study would impact the safety of the individual participant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Complete wound clearing of infection | 28 days
  Proportion of subjects with foot ulcer infection completely cleared at or by 28 days of AppliGel-G treatment compared to proportion of subjects with foot ulcer infection completely cleared at or by 28 days of control treatment

SECONDARY OUTCOMES:
Incidence of infection cleared | 28 days
  Incidence of infection cleared at Day 14
DFU Volume % Change | 28 days
  percent change in DFU volume, measured weekly and compared to baseline
DFU Area % Change | 28 days
  percent change in DFU area, measured weekly and compared to baseline

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Georgetown University Hospital Center, Washington D.C., District of Columbia
  - Florida Medical Center & Research, Inc., Miami, Florida
  - GF Professional Research, Corp., Miami Lakes, Florida
  - Advanced Foot and Ankle Institute of Georgia LLC, Smyrna, Georgia
  - Union Memorial Hospital, Baltimore, Maryland
  - Detroit Clinical Research Center, PC, Farmington Hills, Michigan
  - Utah Valley Medical Center, Provo, Utah